CLINICAL TRIAL: NCT00941499
Title: Hepatic Arterial Infusion of Oxaliplatin in Combination With Systemic Fluorouracil, Leucovorin and Bevacizumab With/Without Cetuximab by K-RAS Mutational Status and Liver Function for Advanced Cancers Metastatic to the Liver
Brief Title: Hepatic Arterial Infusion Oxaliplatin + 5FU, Leucovorin, and Bevacizumab +/- Cetuximab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0023; NCI-2011-00538 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Liver; Oxaliplatin; Eloxatin; Bevacizumab; Avastin; Anit-VEGF monoclonal antibody; rhuMAb-VEGF; 5-fluorouracil; 5-FU; Adrucil; Efudex; Leucovorin; Citrovorum; Wellcovorin; Cetuximab; C225; Erbitux; IMC-C225
MeSH Terms: interventions — Oxaliplatin; Fluorouracil; Bevacizumab; Cetuximab; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): HAI oxaliplatin in combination with HAI 5-fluorouracil and IV bevacizumab
  Interventions: Drug: HAI Oxaliplatin; Drug: 5-FU; Drug: Bevacizumab
- Group 2 (Experimental): HAI oxaliplatin in combination with IV 5-fluorouracil, leucovorin, bevacizumab, and cetuximab
  Interventions: Drug: HAI Oxaliplatin; Drug: Bevacizumab; Drug: Leucovorin; Drug: 5-FU
- Group 3 (Experimental): HAI oxaliplatin in combination with IV bevacizumab.
  Interventions: Drug: HAI Oxaliplatin; Drug: Bevacizumab
- Group 4 (Experimental): HAI oxaliplatin in combination with IV bevacizumab and cetuximab.
  Interventions: Drug: HAI Oxaliplatin; Drug: Cetuximab; Drug: Bevacizumab

INTERVENTIONS:
Drug: HAI Oxaliplatin — 140 mg/m^2 by HAI (hepatic arterial infusion)over 2 hours on Day 1 of each 21 day cycle
  Other Names: Eloxatin
Drug: 5-FU — 900-1750 mg/m^2 HAI infusion over 24 hours on Days 1 - 2 of each 21 day cycle.
  Other Names: 5-Fluorouracil; Adrucil; Efudex
  Arms: Group 1
Drug: Bevacizumab — 10 mg/Kg by vein on Day 1 of 21 day cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
  Arms: Group 1; Group 2; Group 3
Drug: Cetuximab — Loading dose of 250-500mg/m^2 and Maintenance dose of 125-250 mg/m^2 by vein on Day 1 of 21 day cycle.
  Other Names: C225; Erbitux; IMC-C225
  Arms: Group 4
Drug: Leucovorin — 200 mg/m^2 by vein on Days 1 and 2 of each 21 day cycle.
  Other Names: Citrovorum; Wellcovorin
  Arms: Group 2
Drug: 5-FU — 300-400 mg/m^2 bolus + 600-1000 mg/m^2 infusion over 22 hours on Days 1-2 of each cycle.
  Other Names: 5-Fluorouracil; Adrucil; Efudex
  Arms: Group 2
Drug: Bevacizumab — 7.5 - 15 mg/Kg by vein on Day 1 of 21 day cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
  Arms: Group 4

SUMMARY:
The goal of this clinical research study is to find the best combination of oxaliplatin, bevacizumab, 5-fluorouracil, leucovorin, and cetuximab that can be given to patients with advanced cancer that has spread to the liver. Different combinations of these drugs will be used, and the safety of all drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Oxaliplatin is designed to keep new cancer cells from growing.

5-fluorouracil is designed to block the way cancer cells grow and divide, which may slow or stop their growth and keep them from spreading throughout the body. This may cause the cancer cells to die.

Leucovorin is designed to strengthen the effect of 5-fluorouracil by reducing tumor cell resistance to 5-fluorouracil. BECAUSE OF A PHARMACY SHORTAGE OF IV LEUCOVORIN, PATIENTS WILL CONTINUE TREATMENT WITHOUT LEUCOVORIN UNTIL IT BECOMES AVAILABLE.

Bevacizumab is designed to block the growth of blood vessels that supply nutrients necessary for tumor growth. This may prevent or slow down the growth of cancer cells. Bevacizumab is no longer FDA approved to treat breast cancer.

Cetuximab is designed to prevent or slow down the growth of cancer cells by blocking proteins inside the cancer cell, called the epidermal growth factor receptor (EGFR).

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study "arm" (group) based on the results of your screening tests. All patients will receive oxaliplatin and bevacizumab. If your doctor thinks it is in your best interest, you will also receive cetuximab. However, recent studies have found that cetuximab, when given alone or in combination with other chemotherapy drugs, was not effective when given to patients with colorectal cancer that had a K-RAS mutation. If you have colorectal cancer and you are tested for and do not have the K-RAS gene, you will also receive cetuximab. Patients with normal liver function will also receive 5-FU.

* If you are in Arm A, you will receive oxaliplatin, 5-FU, and bevacizumab.
* If you are in Arm B, you will receive oxaliplatin, 5-FU, leucovorin, bevacizumab, and cetuximab.
* If you are in Arm C, you will receive oxaliplatin and bevacizumab.
* If you are in Arm D, you will receive oxaliplatin, bevacizumab, and cetuximab.

Arm A:

All participants will receive the same dose levels of oxaliplatin and bevacizumab.

You will be assigned to a dose level of 5-FU based on when you joined this study. Up to 4 dose levels of 5-FU will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen.

Arm B:

All participants will receive the same dose levels of oxaliplatin, bevacizumab, and leucovorin.

You will be assigned to a combination dose level of 5-FU and cetuximab based on when you joined this study. Up to 4 combination dose levels of 5-FU and cetuximab will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen.

Arm C:

All participants will receive the same dose levels of oxaliplatin.

You will be assigned to a dose level of bevacizumab based on when you joined this study. Up to 4 dose levels of bevacizumab will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen.

Arm D:

All participants will receive the same dose levels of oxaliplatin.

You will be assigned to a combination dose level of bevacizumab and cetuximab based on when you joined this study. Up to 4 combination dose levels of bevacizumab and cetuximab will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen.

In each group, after the highest tolerable dose of the study drug combination is found, up to 12 additional patients will receive that dose level.

Additionally, for Arm A and Arm B, after the highest tolerable dose of the study drug combination is found, up to 20 additional participants with colorectal cancer will be added to Arm A and Arm B.

Catheter Placement for Study Drug Administration:

You will be hospitalized to receive the study drug combination. On the day of your admission to the hospital, you will have a catheter (a sterile flexible tube that will be placed in the hepatic artery [a blood vessel in the liver] while you are under local anesthesia) through which you will receive the study drugs. The catheter will be placed and removed during each cycle. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

You must lay in bed for the entire time that the catheter is in place. In some cases, the catheter will be removed right after your chemotherapy is complete. In some cases, the catheter may remain in overnight. Therefore, you must remain in bed until the catheter is removed.

Study Drug Administration:

Arm A:

On day 1 of each 21 day cycle you will receive oxaliplatin through the hepatic arterial catheter over 2 hours. You will then receive 5-FU over 24 hours through the hepatic arterial catheter. You will then receive bevacizumab by vein over 1 1/2 hours.

Arm B:

On day 1 of each 21 day cycle you will receive oxaliplatin through the hepatic arterial catheter over 2 hours and 5-FU and leucovorin by vein over 24 hours on Days 1 and 2 of each cycle (a total of 48 hours). You will then receive bevacizumab by vein over about 1 1/2 hours, followed by cetuximab by vein over 1-2 hours.

Arm C:

On day 1 of each 21 day cycle you will receive oxaliplatin through the hepatic arterial catheter over 2 hours and bevacizumab by vein over about 1 1/2 hours.

Arm D:

On day 1 of each 21 day cycle you will receive oxaliplatin through the hepatic arterial catheter over 2 hours and you will receive bevacizumab by vein over about 1 1/2 hours. You will also receive cetuximab by vein over about 1-2 hours on Day 1 of each cycle.

Study Visits:

At each study visit, you will be asked about any other drugs you may be receiving and about any side effects you may be having.

On Day 1 of Cycle 1:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be used to test your blood's ability to clot.
* If your study doctor thinks it is needed, you will have an ECG.
* Women who are able to become pregnant will have a urine pregnancy test.

On Day 2 of Cycle 1:

-You will have a physical exam, including measurement of your weight and vital signs.

On Day 1 of Cycles 2 and beyond:

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* If your study doctor thinks it is needed, you will have an ECG.
* Women who are able to become pregnant will have a urine pregnancy test.

On Day 2 of Cycles 2 and beyond:

-You will have a physical exam, including measurement of your weight and vital signs.

At the end of each cycle, blood (about 1 teaspoon) will be drawn to test your blood's ability to clot.

At the end of Cycle 2 and then every 2-3 cycles after that, you will have scans to check the status of the disease. This may include a chest x-ray, CT scan, MRI scan, a PET scan and/or a PET/CT scan. If the study doctor thinks it is more appropriate for you, other types of scans may need to be performed. The study doctor will discuss these scans with you, and you may be asked to sign a separate consent form.

Length of Study:

You may continue to receive the study drug combination for as long as you are benefitting. You will be taken off study if the disease gets worse or if you experience any intolerable side effects.

Follow-Up:

About 6 weeks after your last dose of study drugs, the following tests and procedures will be performed:

* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have a physical exam, including measurement of your weight and vital signs.

This is an investigational study. All of the study drugs are FDA-approved and commercially available for use in other types of cancer:

* 5-FU - for cancers of the breast, pancreas, colon/rectum, stomach, and a type of skin cancer (superficial basal cell carcinoma).
* Oxaliplatin and leucovorin - for colorectal cancer.
* Bevacizumab - for colorectal and lung cancers.
* Cetuximab - for colorectal and head/neck cancers.

It is investigational to give the study drugs together for advanced cancer.

Up to 198 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed cancer with metastatic liver metastases.
2. Patients should be refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that increases survival by at least 3 months, unless the drugs in the protocol regimen are part of the standard of care.
3. Performance status Eastern Cooperative Oncology Group (ECOG) 0-2 (Capable of all self care but unable to carry out any work activities). Pediatric: performance status Karnovsky (>10) or Lansky (<10).
4. Adequate renal function (Serum Creatinine </= 2.0 mg/dL). Pediatric: serum creatinine </= 1.5 mg/dL or 2x upper limit of normal, for age.
5. Patients will be stratified by liver function tests: Normal liver function: Total Bilirubin </= 3 mg/dL, Alanine aminotransferase (ALT) </= 5 times upper normal reference value. Abnormal liver function: Total bilirubin >3 mg/dL and/or elevated ALT > 5 x upper limit of normal (ULN). If bilirubin is >/= 5 mg/dL, fluorouracil (5FU) dose will be omitted. Both of the above groups will be eligible.
6. Adequate bone marrow function (Absolute Neutrophil Count (ANC) >/=1500 cells/uL; Platelets (PLT) >/= 100,000 cells/uL).
7. At least three weeks from previous cytotoxic chemotherapy before day 1 of hepatic arterial infusion (HAI) infusion. After targeted or biologic therapy, there should be 5 half-lives or three weeks, whichever is shorter.
8. All females in childbearing age MUST have a negative urine human chorionic gonadotropin (HCG) test unless prior hysterectomy or menopause (defined as age above 55 and six months without menstrual activity). Patients should not become pregnant or breast feed while on this study. Sexually active patients should use effective birth control.
9. Ability to sign informed consent form. Pediatric: age 7-18 would sign assent, (<7 would not assent), parent or guardian would sign consent.
10. Patients with colorectal cancer must agree to K-RAS mutational status screening, if not available. If tissue is not available, patients can enter on trial, but not on the cetuximab arms.

Exclusion Criteria:

1. Pregnant females.
2. Inability to complete informed consent process and adhere to protocol treatment plan and follow-up requirements.
3. Serious or non-healing wound, ulcer or bone fracture.
4. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days.
5. Uncontrolled systemic vascular hypertension (Systolic blood pressure > 140 mmHg, Diastolic Blood Pressure > 90 mmHg).
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parental antibiotics, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patients already in uncompensated liver failure (i.e. Child Pugh Liver Classification C).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Dose Limiting Toxicity (DLT) of Intra-Arterial Hepatic Oxaliplatin | 21 days
  If more than 33% of patients enrolled in any particular dose level develop DLT, the treatment will continue at the dose level immediately below. If not more than 33% of the patients in the cohort develop DLT, this cohort will be considered the MTD. DLT defined as any Grade 3 or 4 non-hematologic toxicity as defined in NCI CTC v3.0, any Grade 4 hematologic toxicity lasting at least 3 weeks or longer (as defined by the NCI CTC), despite supportive care or associated with bleeding and/or sepsis; any Grade 4 nausea or vomiting > 5 days despite maximum anti-nausea regimens, and any other Grade 3 non-hematologic toxicity including symptoms/signs of vascular leak or cytokine release syndrome, but excluding alopecia; or any severe or life-threatening complication or abnormality not covered in the NCI CTC. The MTD defined by DLTs that occur in the first cycle.
Anti-Tumor Efficacy | After 2, 21 day cycles
  Response Evaluation Criteria in Solid Tumors (RECIST) guidelines used to assess the efficacy of this regimen. A 20% increase in the sum of the greatest longitudinal diameters considered stable disease in the absence of clinical symptoms. An exploratory analysis of radiographic tool measuring the diameter of tumor lesions and comparing their tissue density in comparison with liver function studies and serum biochemical markers performed among study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD, PHD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org